CLINICAL TRIAL: NCT05173038
Title: Sun Yat-sen Memorial Hospital
Brief Title: Second Ejaculate and IUI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: Second Ejaculate 2021-8-17
Record Dates: First submitted 2021-12-21; First posted 2021-12-29 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy Rate; Sperm Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- second ejaculate group
  Interventions: Behavioral: second ejaculate
- first ejaculate group

INTERVENTIONS:
Behavioral: second ejaculate — group patients received IUI for pregnancy assistance 1 hour after the first sperm extraction. The two semen were mixed and treated.
  Groups: second ejaculate group

SUMMARY:
The WHO operation specification requires men to maintain a 2-7-day ejaculation abstinence period before semen examination, but it does not mention the possibility of obtaining a second sample immediately after the first sample for evaluation, and the significance of the evaluation of the second sample for fertility. There is a certain fluctuation level in sperm concentration detection. Patients with normal previous detection may have lower sperm concentration on the day of IUI, resulting in the trouble of canceling IUI. It is not clear whether patients with previous oligospermia can obtain more sperm with better vitality and improve the success rate of IUI by taking sperm again. Some retrospective studies found that when the semen abstinence period of oligozoospermia men was as short as 40 minutes, the changes of sperm motility and sperm concentration were significantly improved, but there was no difference in the conclusions of other studies. A small number of assisted reproduction studies found that IUI with samples obtained during abstinence period of less than 2 days could obtain better pregnancy rate. However, the quality and sample size of these retrospective studies are limited, the repeatability is not good enough, and the conclusions are still controversial. We designed a randomized controlled study. Semen examination was performed after sperm extraction. If the sperm concentration after treatment was less than 10m, the subjects were included in the study. They were randomly divided into two groups. Group 1 received IUI for pregnancy assistance directly, and group 2 received IUI for pregnancy assistance 1 hour after the first sperm extraction. The two semen were mixed and treated. 205 subjects were included in the two groups. We tried to explore whether secondary sperm extraction in patients with low IUI concentration can improve the success rate of IUI pregnancy.

ELIGIBILITY:
Inclusion Criteria:

- Man

1. Male infertility (primary or secondary infertility)
2. Age 22 ~ 80 years old;
3. Body mass index < 30 kg / m2;
4. Normal levels of FSH, LH, t and PRL;
5. Semen concentration and vitality were normal or slightly abnormal (TSC ≥ 10 million / ml, PR ≥ 20%, vitality ≥ 30%), which was consistent with the indication of IUI assisted pregnancy;
6. On the day of IUI, the male side took the semen and the TSC was less than 10m / ml

Women's standard

1. Age 20 ~ 40 years old
2. Body mass index < 30 kg / m2;

3）FSH<10U/L、AMH>1.1ng/ml

4) Bilateral fallopian tubes are unobstructed

Exclusion Criteria:

* Man

It has performed vasectomy, orchitis, unilateral orchiectomy, ejaculation difficulty, retrograde ejaculation, diabetes, cardiovascular disease, drug treatment of psychological or genetic diseases.

Woman

1. Previous history of intrauterine adhesion;
2. Hydrosalpinx;
3. B-ultrasound suggests that endometriosis cyst may be;

Ages: 22 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: patient who come to sun yat-sen memorial hospital to do IUI
Sampling Method: Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pregnacy rate | 2021-8-20~2024.12.30

SECONDARY OUTCOMES:
Semen concentration | 2021-8-20~2024.12.30
semen volume | 2021-8-20~2024.12.30
forward movement rate | 2021-8-20~2024.12.30
non forward movement rate | 2021-8-20~2024.12.30
proportion of immobile sperm | 2021-8-20~2024.12.30
total number of motile sperm after treatment. | 2021-8-20~2024.12.30
Abortion rate | 2021-8-20~2024.12.30

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No